CLINICAL TRIAL: NCT07003217
Title: The Effects of Virtual Reality-Based Practical Education on Learning Satisfaction, Technology Acceptance, Learning Motivation, and Learning Achievement of Physical Therapy Students
Brief Title: The Effects of Virtual Reality-Based Practical Training on Physical Therapy Students
Acronym: VR-STAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hyoshil Yoon, Ph.D. Student and Principal Investigator, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HY-VRPT-001; SYU 2024-02-022-002 (Other: Sahmyook University Institutional Review Board (IRB))
Record Dates: First submitted 2025-05-01; First posted 2025-06-04 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers - Male and Female
Keywords: virtual reality; learning satisfaction; technology acceptance; learning motivation; learning achievement

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were unaware of their group assignment (VR-based or video-based education) to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality-based practical education (Experimental): Before the start of the experiment, the participants in the experimental group were provided with instructions on the usage and safety precautions of the head-mounted display (HMD; Pico 4 Enterprise, Pico Technology, China, 2022). All participants were given a disposable facial hygiene cover for the HMD to ensure hygienic use, and those who wore glasses were also instructed on how to properly wear the device.
  Each participant adjusted the HMD to fit their head size and used hand controllers to sequentially select and perform four target musculoskeletal special tests: the Pronator Teres Test, Hawkins-Kennedy Test, Yergason's Test, and Neer's Test. Each VR video lasted approximately 3 to 4 minutes and was designed to allow 180° rotation. Participants engaged in the VR training once per day.
  After the session, post-tests were conducted to assess learning satisfaction, technology acceptance, learning motivation, and learning achievement.
  Interventions: Behavioral: Virtual Reality-based practical education
- Video Watching-based practical education (Active Comparator): The control group received the same musculoskeletal special test content through traditional video-watching instruction. The participants watched the videos while seated individually in a laboratory at S University. Each video lasted approximately 3 to 4 minutes, and the training was conducted once per day.
  Pre- and post-tests were administered to evaluate learning satisfaction, technology acceptance, learning motivation, and learning achievement.
  Interventions: Behavioral: Video Watching-based practical education

INTERVENTIONS:
Behavioral: Virtual Reality-based practical education — VR-based practical education is an interactive learning method that utilizes virtual reality, where participants engage in a 3D environment for learning.
  Arms: Virtual Reality-based practical education
Behavioral: Video Watching-based practical education — Video Watching-based practical education is a passive learning method, where information is delivered solely through video viewing.
  Arms: Video Watching-based practical education

SUMMARY:
The purpose of this study is to investigate the effects of virtual reality (VR)-based education and video watching-based education on physical therapy students' learning satisfaction, technology acceptance, learning motivation, and learning achievement during musculoskeletal special test training. As technology continues to evolve, tech-assisted learning has emerged as a notable approach in modern education. Among these technologies, VR has gained significant attention for its ability to provide immersive and interactive learning environments for both educators and students. VR applications have expanded into the medical field and are increasingly integrated into health science education. Recently, VR tools have moved beyond desktop-based systems to more accessible platforms like mobile apps and head-mounted displays. In medical education, 3D environments enable engaging and self-directed learning that helps learners understand anatomical structures and build confidence in practical skills. In physical therapy, practical education is important, as therapists must accurately choose and perform special tests. Studies suggest that VR-based training is effective in practical education in physical therapy. Although VR has been applied in rehabilitation for stroke and osteoarthritis patients, VR-based educational research targeting undergraduate physical therapy students is lacking. This study hypothesizes that VR-based practical education is more effective than traditional video watching-based education in improving students' learning satisfaction, technology acceptance, learning motivation, and learning achievement. Participants will be randomly assigned to a VR-based experimental group or a video watching-based control group.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the effects of virtual reality (VR)-based practical education for college students in the department of physical therapy on learning satisfaction, technology acceptance, learning motivation, and learning achievement. The four specialized musculoskeletal tests were the pronator teres test, Hawkins Kennedy test, Yergason's test, and Neer's test. The participants of this study were students from the department of physical therapy at S University in Seoul, South Korea, and were classified into 28 participants in the experimental group using VR-based practical education and 24 participants in the control group using video watching-based practical education through random assignment. Both groups participated in the study for the same period of 1 day, a total of 1 time, for 10 to 15 minutes. When selecting participants for the study, a simulator sickness questionnaire (SSQ) was conducted along with general characteristics to evaluate the symptoms of motion sickness, and one or more of the 16 items were excluded from the study if they were at a 'severe level'. Pre- and post-surveys were administered on learning satisfaction, technology acceptance, learning motivation, and learning achievement.

ELIGIBILITY:
Inclusion Criteria:

* students enrolled in the Department of Physical Therapy at S University in Seoul, South Korea
* individuals who had received prior instruction on the four tests included in the study
* those who did not report any of the 16 SSQ items at the "severe" symptom level
* those who fully understood the purpose and procedures of the study and agreed to participate by providing informed consent.

Exclusion Criteria:

* Individuals who have not learned about the four tests included in the study
* those with health issues that limit the use of VR equipment
* those who do not consent to participate in the study
* those who report 'severe' symptoms on any of the 16 items of the Simulator Sickness Questionnaire (SSQ)
* individuals with disabilities, or pregnant women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Learning Satisfaction | Immediately before and after intervention
  The learning satisfaction scale consists of 19 items in total and is divided into three parts. It consists of three items on experience with the system, seven items on feelings about the system, and nine items on satisfaction with the learning approach. The reliability of the learning satisfaction survey used in this experiment is .91 with a cronbach 's α value.
  The learning satisfaction survey items were composed of a 7-point Likert scale.

SECONDARY OUTCOMES:
Technology Acceptance | Immediately before and after intervention
  Technology acceptance consists of usefulness and ease of use of VR educational technology, and the questionnaire consists of 6 and 7 questions, respectively, for a total of 13 questions. The reliability is Cronbach 's α value of .95 for usefulness and .94 for ease of use. The technology acceptance questionnaire items consisted of a 7-point Likert scale.
Learning Motivation | Immediately before and after intervention
  Learning motivation was designed as a questionnaire with reference to previous studies. It consists of a total of 7 items , including questions about the importance and value of the topic. The items were reorganized to be appropriate for this study with reference to previous papers. The reliability is .79 with Cronbach 's α value. The learning motivation questionnaire items were designed on a 7-point Likert scale.
Learning Achievement | Immediately before and after intervention
  Learning achievement was assessed by a 12-item quiz to assess students' understanding of academics. The quiz items were validated by a doctoral degree holder and an educational expert with extensive experience in physical therapy practice education. The pre- and post-tests of learning achievement consisted of the same items.
  Participants were undergraduate students in the Department of Physical Therapy who had studied four musculoskeletal special tests: the Pronator Teres Test, the Hawkins-Kennedy Test, the Yergason's Test, and the Neer 's Test. They were given three questions on each test. The 12 questions on the learning achievement quiz consisted of short answer or multiple choice questions.

CONTACTS AND LOCATIONS:
Overall Officials: Hyoshil Yoon, Ph.D. Candidate, Principal Investigator — Sahmyook University
Locations (1):
- Sahmyook University, Seoul, Dongdaemoon-gu, South Korea

IPD SHARING:
Plan to Share IPD: No
The research results will be published through a journal.